CLINICAL TRIAL: NCT03637751
Title: Temporal Genomics Mechanisms Underlying Disease and Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Idan Shalev, Assistant Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1R21AG055621-01A1 (NIH)
Record Dates: First submitted 2018-08-16; First posted 2018-08-20 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Gene Expression in Response to Acute Stress

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental design (Experimental): Testing will be carried out in Penn State's Clinical Research Center (CRC). The CRC has rooms for conducting the Trier Social Stress Test (TSST) stress-task and for resting. Participants will make two visits to the CRC, one week apart, on the same day of the weekday. Sessions will be scheduled from 11:00 am to 4:15 pm. We will use a randomized counter-balanced order for the two sessions (i.e., TSST and control conditions) with group membership blind to the subjects and lab personnel.
  Interventions: Behavioral: Behavioral
- Control design (Experimental): In the no-stress control condition, participants will be instructed to sit in a room, read magazines, and to refrain from any stressful activities (e.g., cell-phone use will be restricted).
  Interventions: Behavioral: Control condition

INTERVENTIONS:
Behavioral: Behavioral — Trier Social Stress Test
  Arms: Experimental design
Behavioral: Control condition — In the no-stress control condition, participants will be instructed to sit in a room, read magazines, and to refrain from any stressful activities (e.g., cell-phone use will be restricted).
  Arms: Control design

SUMMARY:
Given the salient role of early-life adversity and the resulting biological embedding in disease risk, there is a critical need to understand the mechanisms operating at multiple levels of analysis in order to promote effective clinical treatments and intervention efforts for survivors. An example for such an effort could be to utilize models of dynamic cellular markers as individual-level factors to account for variation in intervention response and clinical outcomes. Results of this study will lead to new knowledge about specific gene expression pathways in response to stress, and whether the response is moderated by previous exposure to early adversity, shorter telomere length (a marker of cellular aging) and self-report mental-health measures. Thus, the long-term effects of this study will advance our understanding on stress-related transcriptomic changes that play a downstream role in disease susceptibility and accelerated aging, with the goal of targeting specific pathways and genes for potential intervention studies and pharmacological treatments to reverse the effects of exposure to early adversity. For example, considering high failure rates for depression treatments, and in order to tailor individual interventions, identifying objective changes in stress-induced gene expression may help to predict intervention efficacy in clinical and non-clinical settings, as seen, for example, in breast and leukemia cancers. Thus, findings will have a range of impacts for basic science, intervention studies and clinical practice that will influence treatments to match the specific cellular processes operating within an individual.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25
* Without significant medical illness or endocrine illness (for example, asthma, diabetes, thyroid disease or pituitary gland disorders)
* Currently non-smokers
* Not pregnant and had not given birth in the past year
* Not using medication on a regular basis besides oral contraceptives to allow generalizability to adult women.

Exclusion Criteria:

* Recent infection or illness
* Use of abused drugs
* Immune disease, ascertained during the phone interview.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-08-21 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Gene expression via RNAseq | Gene expression over 5 hours in response to stress or a no-stress condition

CONTACTS AND LOCATIONS:
Locations (1):
- Biobehavioral Health Building, University Park, Pennsylvania, United States